CLINICAL TRIAL: NCT00559169
Title: Study of Verapamil in Refractory Catamenial Epilepsy
Brief Title: Verapamil and Catamenial Epilepsy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: protocol changed and a new study using verapamil in epilepsy will be started in the near future
Sponsor: University Health Network, Toronto (Other)
Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UHN-TWH-VER-001
Record Dates: First submitted 2007-11-14; First posted 2007-11-16 (Estimated); Last update posted 2010-04-08 (Estimated); Status verified 2007-11

CONDITIONS: Catamenial Epilepsy
Keywords: epilepsy; seizures; menstrual cycle
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Verapamil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: verapamil hyrochloride — 80 mg daily by mouth, 5 days prior to menses for 3 months
  Other Names: apo-verap, isoptin

SUMMARY:
One in 3 epilepsy patients have refractory seizures. This drug resistance is likely related to the over expression of multidrug resistance proteins (MDR). Progesterone is a known inhibitor of MDRs and the low level of this hormone during the menstrual cycle may exacerbate seizures, perhaps explaining catamenial epilepsy; i.e. seizures occurring during the menstrual cycle. Verapamil suppresses seizures in animal models of epilepsy perhaps by inhibiting MDRs and thus may help patients with refractory seizures. If the study shows improved seizure control, the results will help establish the role of MDRs in refractory epilepsy.

ELIGIBILITY:
Inclusion Criteria:

* females
* at least 2 seizures per month
* more than 50% of the seizures occur 7 days before or 7 days after the onset of menses
* patient of the Toronto Western Hospital Epilepsy Clinic

Exclusion Criteria:

* cardiovascular history

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2009-02; Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
the percent reduction in seizure frequency | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Danielle Andrade, MD, Principal Investigator — College of Physicians and Surgeons of Ontario
Locations (1):
- Toronto Western Hospital, Toronto, Ontario, Canada